CLINICAL TRIAL: NCT01829516
Title: The Effects of Intranasal Oxytocin on Social Cognition, Implicit Preferences and Craving in Moderate to Heavy Social Alcohol Drinkers
Brief Title: Intranasal Oxytocin and Social Cognition, Implicit Preferences and Craving in Alcohol Drinkers
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Principal Investigator, Jennifer Mitchell, Principal Investigator, University of California, San Francisco
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: Oxytocin
Record Dates: First submitted 2013-04-09; First posted 2013-04-11 (Estimated); Results first posted 2016-06-27 (Estimated); Last update posted 2016-07-27 (Estimated); Status verified 2016-06

CONDITIONS: AOD Use, Abuse, and Dependence
MeSH Terms: interventions — Oxytocin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Oxytocin (Experimental): 50 moderate to heavy social alcohol users will receive a single dose 40 IU of intranasal oxytocin.
  Interventions: Drug: Oxytocin
- Placebo (Placebo Comparator): 50 moderate to heavy social alcohol users will receive a single dose 40 IU of intranasal placebo.
  NOTE: This is a cross-over design and subjects will participate in both arms.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Oxytocin — Intranasal oxytocin
  Other Names: Syntocinon
  Arms: Oxytocin
Drug: Placebo — Intranasal placebo
  Arms: Placebo

SUMMARY:
This is a randomized, placebo controlled, double blind crossover study of the effects of intranasal oxytocin on social cognition, implicit preferences and craving in moderate to heavy social alcohol drinkers.

DETAILED DESCRIPTION:
Impaired social functioning is an important feature of substance use disorders. Social deficits are a risk factor for developing substance use disorders as well as a consequence of substance abuse. Improved social functioning is also a key goal of effective substance abuse treatments. While treatment of disrupted social networks is a mainstay of psychosocial substance abuse treatments, there are currently no pharmacological interventions aimed at improving social functioning in individuals with substance use disorders. Oxytocin administration may shift preference from substance related cues to social cues and may decrease subjective craving for alcohol.

The specific aims are:

1. To examine the effects of intranasal oxytocin administration on social cognition in moderate to heavy social alcohol drinkers.
2. To examine the effects of intranasal oxytocin administration on alcohol craving.
3. To examine the effects of intranasal oxytocin administration on implicit preferences for drug-related and social stimuli in moderate to heavy social alcohol drinkers.

ELIGIBILITY:
Inclusion Criteria:

* Subject is a volunteer between 18 and 50 years of age.
* If female, subject is non-lactating, not pregnant, and using a reliable contraception method (i.e. abstinence, intrauterine device [IUD], hormonal birth control, or barrier method).
* Subject is able to read and speak English.
* Subject is able and willing to provide written informed consent.
* Subject is able to understand and follow the instructions of the investigator and understand all screening questionnaires.
* Subject is in good health.

Exclusion Criteria:

* Positive urine drug screen (except marijuana).
* Using cocaine, stimulants (other than nicotine and caffeine), amphetamines, hallucinogens, ecstasy, opiates, sedatives, pain pills, sleeping pills, or other psychoactive drugs within 2 weeks of the start of the study (except marijuana) OR more than 10 times in the last year (except marijuana).
* Marijuana use more than 3 times/week.
* Has a current dependence on, or addiction to any psychoactive drug (except nicotine or caffeine) including alcohol OR a recent history of substance abuse other than alcohol, tobacco or marijuana.
* Clinically significant medical or psychiatric illness requiring treatment as determined by screening blood tests, medical history, and/or physical exam performed or reviewed by the study physician.
* BAC level > 0.05% at the beginning of screening visit (within margin of error of detection).
* Has a neurological dysfunction or psychiatric disorder (confirm with study physician).
* Has a history of brain trauma (confirm with study physician).
* Has an allergy or intolerance to oxytocin.
* Subject has received an investigational drug within 30 days of Screening Visit.
* Subject is considered unsuitable for the study in the opinion of the investigator, nurse practitioner, or study physician for any other reason.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2013-05; Primary Completion 2014-05 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Josh Woolley, MD, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- Ernest Gallo Clinic and Research Center, Emeryville, California, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Sixty-one nontreatment-seeking subjects were recruited online. Eligible subjects met DSM-IV criteria for alcohol abuse, but were excluded if physically dependent on alcohol. These subjects were screened to yield 39 eligible subjects. Of the 39 subjects deemed eligible, 7 did not return after the screening visit, resulting in 32 enrolled subjects.
Groups:
- Oxytocin First, Then Placebo: 18 moderate to heavy social alcohol users received a single dose 40 IU of intranasal oxytocin followed by a single dose 40 IU of intranasal placebo.
  NOTE: This is a cross-over design and subjects will participate in both arms.
- Placebo First Then Oxytocin: 14 moderate to heavy social alcohol users received a single dose 40 IU of intranasal placebo followed by a single dose 40 IU of intranasal oxytocin.
  NOTE: This is a cross-over design and subjects will participate in both arms.
Period: First Intervention
Arm/Group | Oxytocin First, Then Placebo | Placebo First Then Oxytocin
Started | 18 | 14
Completed | 18 | 14
Not Completed | 0 | 0
Period: Washout Period - 1 Week
Arm/Group | Oxytocin First, Then Placebo | Placebo First Then Oxytocin
Started | 18 | 14
Completed | 18 | 14
Not Completed | 0 | 0
Period: 2nd Intervention
Arm/Group | Oxytocin First, Then Placebo | Placebo First Then Oxytocin
Started | 18 | 14
Completed | 18 | 14
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: This is a crossover study of 39 moderate to heavy social alcohol users who will receive a single dose 40 IU of intranasal oxytocin followed by 40 IU of placebo or vice versa.
Arm/Group | All Study Participants
Number analyzed (Participants) | 39
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 39
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 24

OUTCOME MEASURES:

1. Primary Outcome: Change in Craving on the Alcohol Urge Questionnaire (AUQ) After Administration of Oxytocin vs. Placebo During the 3-week Study.
Description: Change in craving represented by the mean difference in Alcohol Urge Questionnaire (AUQ) craving scores between alcohol and water cues (e.g., a positive alcohol-water score indicates cue-induced craving) after administration of oxytocin vs. placebo during the 3-week study. Craving for alcohol was assessed prior to the water and alcohol cues and again after each stimulus presentation using the 8-item Alcohol Urge Questionnaire (AUQ) (Bohn et al., 1995), in which subjects indicate how much they agree or disagree with statements regarding their alcohol craving on a 7-point Likert scale. AUQ craving scores are calculated by averaging responses to the 8 items. Each item is scored on a 1 to 7 scale (Strongly Disagree = 1 and Strongly Agree = 7). Items 2 and 7 are reverse scored. A total score is computed by averaging the item scores and ranges from 1 to 7. Higher scores reflect greater craving.
Time Frame: Measured just prior to and after each of the water and alcohol cues at visits 2 and 3.
Population: In this crossover study a total of 32 participants were analyzed for each intervention.
Measure: Mean (Standard Error); unit: units on a 7-pt Likert Scale
Groups:
- Oxytocin: 18 moderate to heavy social alcohol users received 40 IU of intranasal oxytocin followed by 40 IU of intranasal placebo and 14 received 40 IU of intranasal placebo first followed by 40 IU of intranasal oxytocin, for a total of 32 participants analyzed.
- Placebo: 14 moderate to heavy social alcohol users received 40 IU of intranasal placebo followed by 40 IU of intranasal oxytocin and 18 received 40 IU of intranasal oxytocin first followed by 40 IU of intranasal placebo, for a total of 32 participants analyzed.
Arm/Group | Oxytocin | Placebo
Number analyzed (Participants) | 32 | 32
units on a 7-pt Likert Scale | 1.11 (0.20) | 0.69 (0.17)

2. Secondary Outcome: Average Percentage of Correct Responses on a Social Perception Task, Reading the Mind in the Eyes Test (RMET) After Administration of Oxytocin vs. Placebo During the 3-week Study.
Description: We will examine the effects of intranasal oxytocin administration on overall RMET performance in moderate to heavy social alcohol drinkers after placebo or oxytocin administration. The RMET has 28 items. Each item is an cropped photo of a person's eyes with four emotion labels around it. The subjects are asked to select which one of the four emotion words best describes the emotion that the eyes are showing. RMET is scored by adding up the total number of correct responses (range 0-28). The mean percent correct is then calculated.
Time Frame: Administered at visits 2 and 3
Population: 1 subject did not complete the RMET task, so only 31 participant responses were analyzed for this task.
Measure: Mean (Standard Error); unit: Mean percent correct responses
Groups:
- Oxytocin; Placebo: In this crossover study, 18 moderate to heavy social alcohol users will receive a single dose 40 IU of intranasal oxytocin followed by a single dose of 40 IU of intranasal placebo and 14 moderate to heavy social alcohol users will receive a single dose 40 IU of intranasal placebo followed by 40 IU of intranasal oxytocin, for a total of 32 completed participants.
Arm/Group | Oxytocin | Placebo
Number analyzed (Participants) | 31 | 31
Mean percent correct responses | 77.2 (1.7) | 76.4 (1.5)

ADVERSE EVENTS:
Time Frame: Over course of 3 week study
Groups:
- Oxytocin: 50 moderate to heavy social alcohol users will receive a single dose 40 IU of intranasal oxytocin.
  Oxytocin
- Placebo: 50 moderate to heavy social alcohol users will receive a single dose 40 IU of intranasal placebo.
  NOTE: This is a cross-over design and subjects will participate in both arms.
  Placebo
Arm/Group | Oxytocin | Placebo
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/32
Other Adverse Events (participants affected / at risk) | 0/32 | 0/32

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes